CLINICAL TRIAL: NCT04470869
Title: Impact of the Psychiatric Intervention OLAF on the Post Traumatic Disorder in the Relatives of Patients Hospitalized in Intensive Care Unit During the SARS-Cov-2 Pandemic Confinement in France.
Brief Title: Impact on the OLAF Intervention to Prevent Post Traumatic Disorders During the Confinement.
Acronym: OLAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: RC31/20/0190
Record Dates: First submitted 2020-07-03; First posted 2020-07-14 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: intensive care unit; confinement; SARS-CoV-2; post-traumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: In this study we aimed to investigated the impact of this intervention to prevent the PTSD in the relatives by comparing the PTSD prevalence in a group of relatives that loved ones were hospitalized after the confinement measure but before the OLAF intervention and a group of relatives that loved ones were hospitalized during the OLAF intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OLAF group (Experimental): The interventional group (OLAF) benefit from a psychiatric follow up, from virtual visiting of the patient and video interview with ICU team.
  Interventions: Other: Phone call
- Control (Placebo Comparator): The control group contains the relatives of patients hospitalized after the confinement measure but before the OLAF intervention. This group benefit from phone contact with the ICU team at the admission in ICU then two contact per week minimum to one contact per day maximum during the stay, excepting the specific phone calls associated with favorable or unfavorable evolution.
  Interventions: Other: Phone call

INTERVENTIONS:
Other: Phone call — The relatives of both groups will be contacted by phone one month after the discharge of the ICU of the death, three month after, six month after and twelve month after. During these interviews the PTSD symptoms, the anxiety and depression symptoms, the complicated grief symptoms (in case of death) and the satisfaction about the ICU stay will be collected.

SUMMARY:
The investigators thought that the confinement measure took in France could induce an increase in the post traumatic syndrome in the relative of patient hospitalized in ICU during this period indeed the restricted visit and the limited interaction with ICU team are documented risk factors for PTSD in this population. The investigators designed an intervention in order to prevent the effect of the confinement measures on PTSD in relatives named OLAF. In this research the investigators aimed to study the impact on this intervention on PTSD.

DETAILED DESCRIPTION:
The hospitalization of a relative in an intensive care unit is an important stress factor for his/ her relatives and previous studies demonstrated that 33% post traumatic disorder (PTSD) following the ICU stay of their loved ones. To response to this issue specific approach have been designed to decrease the stress of the relatives named family centered care. Those approaches are based on the interaction between the ICU team and the relatives and included large time for visiting the patient in the ward. In France the restrictive measures (confinement) took to combat the SARS-CoV-2 pandemic from the 17 march 2020 impacted negatively those family centered care approach by prohibiting the visit in ICU and limiting to interaction between ICU team and relatives to phone calls. The investigators thought that this context could have for consequence an increase in relative anxiety and PTSD. The investigators designed a care intervention named OLAF in order to limit the impact of the confinement on relative psychological state. OLAF intervention permits to the two closest relatives of the patient to be contacted by a psychiatrist and could benefit from a specialized follow up. This intervention is completed by the implementation of virtual visits by video conference that were proposed to the relatives as well as video interview with the ICU team. In this study the investigators aimed to investigated the impact of this intervention to prevent the PTSD in the relatives by comparing the PTSD prevalence in a group of relatives that loved ones were hospitalized after the confinement measure but before the OLAF intervention and a group of relatives that loved ones were hospitalized during the OLAF intervention.

The relative will benefit from psychiatric interview 3 months after their loved ones leave the ICU or died to collect information by phone about the confinement situation they experiment, the satisfaction they had about the patient stay in ICU and their anxiety and depression state. Three-month, six month and twelve months after the discharge of the dead the relative information will be collected by phone about PTSD symptoms, anxiety and depression and complicated grief in case of death of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Contact person (defined as the person that bring a support to the patient et with who the patient had close relationship) aged from more than 18 years old of a patient hospitalized during the confinement and the restricted visited during the SARS-CoV2 pandemic. Two contact persons maximum will be included by patient.
* Affiliated to the social security
* Agreed to participated by oral consent

Exclusion Criteria:

* Physical visits permitted by the end of the confinement
* Language barrier
* Sensorial handicap (blindness or deafness) compromising the comprehension of the information
* Legal protection of adults
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
incidence of PTSD observed 6 months after patient's discharge from the intensive care unit | Month 6
  To demonstrate the benefits of a comprehensive family approach (OLAF) on the incidence of PTSD observed in 2 close referents of a patient, 6 months after leaving the intensive care unit, in the context of confinement linked to the SARS pandemic- CoV2.

SECONDARY OUTCOMES:
incidence of PTSD observed 6 months after patient's death in the intensive care unit | Month 6
  The incidence of PTSD 6 months after patient's death in the intensive care unit
PTSD incidence at month 3 | Month 3
  The incidence of PTSD 3 months after the death or discharge from the intensive care unit
PTSD incidence at month 12 | Month 12
  The incidence of PTSD 12 months after the death or discharge from the intensive care unit
Symptoms incidence at month 3 | Month 3
  The incidence of symptoms of anxiety and / or depression 3 months after death or discharge from the intensive care unit
Symptoms incidence at month 6 | Month 6
  The incidence of symptoms of anxiety and / or depression 6 months after death or discharge from the intensive care unit
Symptoms incidence at month 12 | Month 12
  The incidence of symptoms of anxiety and / or depression 12 months after death or discharge from the intensive care unit
incidence of persistent complicated grief at month 3 | Month 3
  The incidence of persistent complicated grief 3 months after death in intensive care
incidence of persistent complicated grief at month 6 | Month 6
  The incidence of persistent complicated grief 6 months after death in intensive care
incidence of persistent complicated grief at month 12 | Month 12
  The incidence of persistent complicated grief 12 months after death in intensive care

CONTACTS AND LOCATIONS:
Overall Officials: Juliette SALLES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, Occitanie, France

REFERENCES:
- [Derived] Raymond V, Aitout C, Ducos G, Coullomb A, Ferre F, Vardon-Bounes F, Riu-Poulenc B, Seguin T, Boukhatem L, Geeraerts T, Minville V, Fourcade O, Birmes P, Arbus C, Silva S, Salles J. Effectiveness of psychiatric support for PTSD among a cohort of relatives of patients hospitalized in an intensive care unit during the French COVID-19 lockdown-The OLAF (Operation Liaison et Aide aux Familles): A quasi-randomized clinical trial. Gen Hosp Psychiatry. 2023 Sep-Oct;84:266-267. doi: 10.1016/j.genhosppsych.2023.06.009. Epub 2023 Jun 21. No abstract available. PMID 37357092